CLINICAL TRIAL: NCT02407405
Title: Phase II Trial of the MEK1/2 Inhibitor Selumetinib (AZD6244 Hydrogen Sulfate in Adults With Neurofibromatosis Type 1 (NF1) and Inoperable Plexiform Neurofibromas
Brief Title: MEK 1/2 Inhibitor Selumetinib (AZD6244 Hydrogen Sulfate) in Adults With Neurofibromatosis Type 1 (NF1) and Inoperable Plexiform Neurofibromas
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160043; 16-C-0043; NCT02644512 (obsolete NCT alias)
Record Dates: First submitted 2015-04-02; First posted 2015-04-03 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10-08

CONDITIONS: Neurofibromatosis 1 (NF1); Plexiform Neurofibromas (PN)
Keywords: Objective Response; pERK inhibition; MEK Inhibition; Biopsy; Volumetric MRI
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform | interventions — AZD 6244

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Selumetinib 50 mg BID daily
  Interventions: Drug: Selumetinib

INTERVENTIONS:
Drug: Selumetinib — orally 50 mg/dose, every 12 hours every day continuously (1 cycle = 28 days)

SUMMARY:
Background:

Neurofibromatosis type 1 (NF1) is a disorder that can cause plexiform neurofibromas (PNs). These are tumors that grow along nerves. Some PNs cause serious health problems. PNs often can t be operated on because of their large size, location, or number. There are no effective treatments known for people with NF1 and PNs. Researchers want to test if the drug selumetinib (AZD6244 hydrogen sulfate) causes PNs to shrink or slows down their growth.

Objectives:

To test if selumetinib helps treat PNs. To test how the body handles selumetinib and how it affects peoples symptoms.

Eligibility:

People ages 18 and older with NF1, with an inoperable PN that causes morbidity or is growing

Design:

Participants will be screened with:

Medical history and physical exam

Blood, urine, and heart tests

Eye exam

MRI: They lie in a machine that takes pictures of the body.

PN biopsy: A small piece of the tumor is removed by a large needle.

Questionnaires

Participants will swallow selumetinib capsules every 12 hours for several 28-day cycles. The capsules are taken with a full glass of water on an empty stomach. Participants may have only water for 2 hours before and 1 hour after each dose.

Participants will keep a drug diary. They will continue taking the drug as long as they tolerate it and their disease doesn t progress.

Participants will have several visits throughout the study. These will include repeats of the screening tests.

Participants will have a final visit after they stop taking selumetinib.

DETAILED DESCRIPTION:
Background:

* Neurofibromatosis 1 (NF1) is an autosomal dominant disorder with an incidence of 1:3500 in the US. One of the cardinal features of NF1 is the development of histologically benign peripheral nerve sheath tumors called plexiform neurofibromas (PN) in 25-40% of individuals with NF1. Unlike discrete neurofibromas, PN grow along the length of nerves and involve multiple branches of a nerve. They are a major source of morbidity, causing disfigurement, impairment of nerve function, pain, and in some cases development of malignant peripheral nerve sheath tumors.
* Selumetinib (AZD6244) is a novel orally bioavailable mitogen activated protein kinase inhibitor, is a specific inhibitor of MEK 1/2, which may mediate anti-tumor effects in PN by inhibition of downstream signaling of Ras. Selumetinib is currently undergoing evaluation in adult cancers and children with brain tumors and NF1-related plexiform neurofibromas.
* In an NCI phase I trial of selumetinib for children and young adults with NF1 and inoperable PN we have observed preliminary activity with PN volume decrease in >50% of patients enrolled. This degree of activity has not been observed in prior trials directed at PN. While preliminary activity has been seen in most patients enrolled to date, in several patients who required >= 1 dose reduction for toxicity, after an initial volume decrease, the PN volumes appear to be increasing slowly, and in one patient a nodular appearing lesion is not responding to selumetinib. These findings suggest that not all PN types may be responsive to selumetinib and that a certain selumetinib tissue concentration may be required for target inhibition and anti-tumor activity.

Objective:

-Determine the objective response rate (PN volume decrease >=20% compared to baseline) to selumetinib in adult patients with inoperable PN.

Eligibility:

* Patients must be at least 18 years of age with a diagnosis of NF1, with an inoperable, measurable PN that causes morbidity or is growing, which is amenable to percutaneous biopsy, and must be willing to undergo two biopsies.
* Up to 10 patients who meet all criteria, but have PN, which cannot be biopsied safely, will be eligible for the treatment portion of the study.
* Patients must have adequate organ function, be able to undergo serial MRI scans and have recovered from acute toxicity of all prior treatment.

Design:

* This is a single site open label phase II study in which all subjects will receive selumetinib orally approximately every 12 hours until patient develops progression of disease, unacceptable toxicity or, in patients with non-progressive, symptomatic PN at enrollment, a maximum of 2 years (unless they experience a partial response, or an improvement in symptoms or function in which case they may continue until progression of disease).
* Selumetinib will be administered at a dose of 50 mg BID on a continuous dosing schedule (1 cycle =28 days), which is the recommended adult dose. A maximum accrual of 35 evaluable patients to meet the primary objective; while a maximum of 60 patients in total may be enrolled to allow for a small number of screen failures, inevaluable patients and up to 10 patients who cannot safely undergo two biopsies of PNs. Enrollment will proceed over approximately 24 months.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have positive genetic testing for NF1 in a CLIA certified laboratory or a diagnosis of NF1 based on clinical NIH consensus criteria of at least one other diagnostic criterion in addition to the presence of a PN. NF1 mutation analysis will be performed on germline DNA. Histologic confirmation of tumor is not necessary in the presence of consistent clinical and imaging findings, but should be considered if malignant transformation of a PN is clinically suspected. Additional criteria are as follows:

  * Six or more cafe-au-lait macules (>=0.5cm in prepubertal subjects or >=1.5 cm in post pubertal subjects)
  * Freckling in axilla or groin
  * Optic glioma
  * Two or more Lisch nodules
  * A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
  * A first-degree relative with NF1
* Measurable disease: Patients must have at least one measurable PN, defined as a lesion of at least 3 cm measured in one dimension. Patients who underwent surgery for resection of a PN are eligible provided the PN was incompletely resected and is measurable as per criteria above. Measurability and suitability for volumetric MRI analysis of the target PN must be confirmed with the NCI POB prior to enrolling a patient. The target PN will be defined as the clinically most relevant PN, which has to be amenable to volumetric MRI analysis. PN will be classified as typical PN versus nodular PN versus solitary nodular PN prior to enrollment
* The PN must be inoperable, defined as a PN that cannot be surgically completely removed without risk for substantial morbidity due to: encasement of or close proximity to vital structures, invasiveness, or high vascularity of the PN. The PN either causes morbidity or it is growing and has the potential to cause morbidity such as (but not limited to): Head and neck lesions that could compromise the airway or great vessels, paraspinal lesions that can cause myelopathy, brachial or lumbar plexus lesions that could cause nerve compression and loss of function, lesions that could result in major deformity (e.g., orbital lesions) or are significantly disfiguring, and lesions of the extremity that cause limb hypertrophy or loss of function or pain. PN growth will be defined as a >=20% increase in PN volume within approximately 3 years prior to enrollment on this trial.
* Patients must have a PN amenable to a percutaneous biopsy to participate in the biopsy portion of this study, and must be willing to undergo pre-, and on treatment tumor biopsies. There should be no contraindication for serial biopsies. NOTE: Up to 10 patients who meet all criteria, but have PN which cannot be biopsied safely, will be eligible for the treatment portion of the study.
* Must be able to undergo serial MRI scans for response evaluation
* Age >=18 years
* ECOG performance status <=2 (Patients who are wheelchair bound because of paralysis secondary to a plexiform neurofibroma should be considered ambulatory when they are up in their wheelchair. Similarly, patients with limited mobility secondary to need for mechanical support (such as an airway PN requiring tracheostomy or CPAP) will also be considered ambulatory for the purpose of the study.)

  --ECOG Performance Status:*
  * Grade/ECOG
  * 0 Fully active, able to carry on all pre-disease performance without restriction
  * 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  * 2 Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours
  * 3 Capable of only limited self-care, confined to bed or chair more than 50% of waking hours
  * 4 Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  * 5 Dead

    * As published in Am. J. Clin. Oncol.: Oken, M.M., Creech, R.H., Tormey, D.C., Horton, J., Davis, T.E., McFadden, E.T., Carbone, P.P.: Toxicity And Response Criteria Of The Eastern Cooperative Oncology Group. Am J Clin Oncol 5:649-655, 1982.
* Patients must have normal organ and marrow function as defined below:

  * Hemoglobin >=10 g/dL (not requiring RBC transfusions)
  * Absolute neutrophil count >=1,500/mcL
  * Platelets >=100,000/mcL (not requiring platelet transfusions)
  * Total bilirubin <=1.5 upper limit of normal (ULN), with the exception of patients with Gilbert Syndrome
  * ALT(SGPT) & AST(SGOT) <=3.0 X ULN
  * Creatinine <=upper limit of normal institutional limits
  * OR
  * Creatinine clearance >=60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Hematologic parameters for patients undergoing biopsy only: Patients should have INR <=1.4 and PTT <=40 seconds (unless due to lupus anticoagulant). In patients not meeting these parameters, clearance by hematology will be required prior to undergoing a biopsy.
* Cardiac Function: Normal ejection fraction (ECHO) >=53% (if a range is given then the upper value of the range will be used) or cardiac MRI; QTcF <=450 msec.
* Ability of subject or Legally Authorized Representative (LAR)) to understand and the willingness to sign a written informed consent document.
* Willingness to avoid excessive sun exposure and use adequate sunscreen protection if sun exposure is anticipated.
* Willingness to avoid the ingestion of grapefruit and Seville oranges (as well as other products containing these fruits, e.g. grapefruit juice or marmalade) during the study.
* Prior therapy: Patients with NF1 will only be eligible if complete tumor resection is not considered to be feasible without substantial risk or morbidity, or if a patient with a surgical option refuses surgery.

  * Since there is no standard effective chemotherapy for patients with NF1 and PN, patients may be treated on this trial without having received prior medical therapy directed at their PN.
  * Since selumetinib is not expected to cause substantial myelosuppression, there will be no limit to number of prior myelosuppressive regimen for PN or other tumor manifestations associated with NF1 such as optic glioma.
  * Patients who have received previous investigational agents or biologic therapy, such as tipifarnib, pirfenidone, Peg-Intron, sorafenib, or other VEGFR inhibitors are eligible for enrollment.
  * Growth factors that support platelet or white cell number or function must not have been administered within the past 7 days and are not permitted while on the study.
  * At least 6 weeks must have elapsed prior to enrollment since the patient received any prior radiation therapy, and no prior radiation therapy should have been directed at the target PN.
  * At least 4 weeks must have elapsed since receiving medical therapy directed at the PN.
  * At least 4 weeks must have elapsed since any surgeries, with evidence of completed wound healing.
  * Patients who received prior medical therapy for their PN must have recovered from the acute toxic effects of all prior therapy to <= grade 1 before entering this study.
* Informed Consent: Diagnostic or laboratory studies performed exclusively to determine eligibility for this trial must only be done after obtaining written informed consent from all patients, which can be accomplished using the screening consent for this protocol. Studies or procedures that were performed for clinical indications (not exclusively to determine eligibility) may be used for screening or baseline values even if the studies were done before informed consent was obtained, if the patient agrees.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents, or have received an investigational agent within the past 30 days.
* May not have a NF1 related tumor such as optic pathway glioma or malignant peripheral nerve sheath tumor, which requires treatment with chemotherapy or surgery.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements. Patients with HIV who have adequate CD4 counts and who have no requirement for antiviral therapy will be eligible.
* Pregnant or breast-feeding females are excluded due to potential risks of fetal and teratogenic adverse events of an investigational agent. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method. Abstinence is an acceptable method of birth control.
* Prior treatment with selumetinib or another specific MEK 1/2 inhibitor.
* Supplementation with vitamin E greater than 100% of the daily recommended dose.
* Inability to swallow capsules, since capsules cannot be crushed or broken.
* Inability to undergo MRI and/or contraindication for MRI examinations following the MRI protocol. Prosthesis or orthopedic or dental braces that would interfere with volumetric analysis of target PN on MRI.
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption.
* Uncontrolled hypertension (despite medical therapy); blood pressure should be <140/90 in accordance with American Heart Association definition of hypertension.
* While not an exclusion criterion, unless clinically indicated, patients should avoid taking other additional non-study medications that may interfere with the study medications. In particular, patients should avoid medications that are known to either induce or inhibit the activity of hepatic microsomal isoenzymes CYP1A2, CYP2C19 and CYP3A4, as this may interfere with the metabolism of selumetinib.
* Known Cardiac Disorder, including:

  * Known inherited coronary disease
  * Symptomatic heart failure (NYHA Class II-IV prior or current cardiomyopathy, or severe valvular heart disease)
  * Current cardiomyopathy
  * Severe valvular heart disease
  * Atrial fibrillation
  * Ejection fraction (ECHO) <53%
  * QTcF >450 msec
* Known Ophthalmologic conditions, such as:

  * Current or past history of central serous retinopathy
  * Current or past history of retinal vein occlusion
  * Known intraocular pressure (IOP) > 21 mmHg (or ULN adjusted by age) or uncontrolled glaucoma (irrespective of IOP). Patients with known glaucoma and increased IOP who do not have meaningful vision (light perception only or no light perception) and are not experiencing pain related to the glaucoma, may be eligible after discussion with the study chair.
  * Subjects with any other significant abnormality on ophthalmic examination should be discussed with the Study Chair for potential eligibility
  * Ophthalmological findings secondary to long-standing optic pathway glioma (such as visual loss, optic nerve pallor or strabismus) or long-standing orbito-temporal PN (such as visual loss, strabismus) will NOT be considered a significant abnormality for the purposes of the study
* Known severe hypersensitivity to selumetinib or any excipient of selumetinib or history of allergic reactions attributed to compounds of similar chemical or biologic composition to selumetinib
* Have had recent major surgery within a minimum of 4 weeks prior to starting study treatment, with the exception of surgical placement for vascular access.
* Have any unresolved chronic toxicity with CTC AE grade >= 2, from previous anti-NF1 therapy, except for alopecia.
* Clinical judgment by the investigator that the patient should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Determine objective response rate | at each response evaluation visit
  Efficacy

SECONDARY OUTCOMES:
Evaluate immune infiltrate of PN and Peripheral blood for circulating tumor cells | Prior to cycle 2 or 3, at time of progression and/or prior to cycle 2 or 3 after dose reduction
  Evaluate immune infiltrate of PN and Peripheral blood for circulating tumor cells
evalaute change in dermal neurofibroma by photography. | Prior to cycle 5, 9, 13, 17, 21, 25 Then after every 12 cycles
  Evalaute change in dermal neurofibroma by photography
determine time to progression and progression free survival | at time of progression
  Time to progression and progression free survival
correlate 3D MRI responses with % target inhibition of pERK in PN biopsies | rior to cycle 5, 9, 13, 17, 21, 25 Then after every 6 cycles
  Correlate 3D MRI responses with % target inhibition of pERK in PN biopsies
compare pERK inhibition in dermal neurofibromas and PN | Prior to cycle 2 or 3, at time of progression and/or prior to cycle 2 or 3 after dose reduction
  Compare pERK inhibition in dermal neurofibromas and PN
characterize effects on pain, quality of life, physical functioning | Prior to cycle 3, 5, 9, 13, Then after every 12 cycles
  Characterize effects on pain, quality of life, physical functioning
Analyze paired biopsies with mechanisms of response and resistance | Prior to cycle 2 or 3, at time of progression and/or prior to cycle 2 or 3 after dose reduction
  Analyze paired biopsies with mechanisms of response and resistance
Analyze bone marrow derived precursor cells and cytokines before and after treatment | Prior to cycle 3, 5, 9, 13
  Analyze bone marrow derived precursor cells and cytokines before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared. All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Requests for all collected IPD data from clinical trials, conducted under a binding collaborative agreement between NCI/DCTD and a pharmaceutical/biotechnology company, that are not under DSMB monitoring must be in compliance with the terms of the binding collaborative agreement and must be approved by NCI/DCTD and the Pharmaceutical Collaborator (i.e., the NCI ETCTN Director in conjunction with the NCI/DCTD Regulatory Affairs Branch).

REFERENCES:
- [Derived] Gross AM, O'Sullivan Coyne G, Dombi E, Tibery C, Herrick WG, Martin S, Angus SP, Shern JF, Rhodes SD, Foster JC, Rubinstein LV, Baldwin A, Davis C, Dixon SAH, Fagan M, Ong MJ, Wolters PL, Tamula MA, Reid O, Sankaran H, Fang F, Govindharajulu JP, Browne AT, Kaplan RN, Heisey K, On TJ, Xuei X, Zhang X, Johnson BC, Parchment RE, Clapp DW, Srivastava AK, Doroshow JH, Chen AP, Widemann BC. Selumetinib in adults with NF1 and inoperable plexiform neurofibroma: a phase 2 trial. Nat Med. 2025 Jan;31(1):105-115. doi: 10.1038/s41591-024-03361-4. Epub 2025 Jan 6. PMID 39762421
- [Derived] Curry BP, Alvarez R, Widemann BC, Johnson M, Agarwal PK, Lehky T, Valera V, Chittiboina P. Robotic Nerve Sheath Tumor Resection With Intraoperative Neuromonitoring: Case Series and Systematic Review. Oper Neurosurg. 2022 Feb 1;22(2):44-50. doi: 10.1227/ONS.0000000000000051. PMID 35007270
- [Derived] Herrick WG, Kilpatrick CL, Hollingshead MG, Esposito D, O'Sullivan Coyne G, Gross AM, Johnson BC, Chen AP, Widemann BC, Doroshow JH, Parchment RE, Srivastava AK. Isoform- and Phosphorylation-specific Multiplexed Quantitative Pharmacodynamics of Drugs Targeting PI3K and MAPK Signaling in Xenograft Models and Clinical Biopsies. Mol Cancer Ther. 2021 Apr;20(4):749-760. doi: 10.1158/1535-7163.MCT-20-0566. Epub 2021 Feb 3. PMID 33536190
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0043.html